CLINICAL TRIAL: NCT01279031
Title: Randomized Comparison of the Abbott WHITESTAR Signature System With Ellips Tranversal Ultrasound vs. the Alcon Infiniti With the Ozil Torsional Handpiece in Phacoemulsification: A Contralaterally-Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Responsible Party: Melissa Earl, CRO
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Abbott2010-Whitestar
Record Dates: First submitted 2011-01-14; First posted 2011-01-19 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Cataracts; Astigmatism
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abbott WHITESTAR Signature System (Experimental): Abbott WHITESTAR Signature System with Ellips Transversal Ultrasound
  Interventions: Device: Abbott WHITESTAR Signature System with Ellips Transversal Ultrasound
- Alcon Infiniti (Experimental): Alcon Infiniti with the OZIL Torsional Handpiece
  Interventions: Device: Alcon Infiniti wiht the OZIL Torsional Handpiece

INTERVENTIONS:
Device: Abbott WHITESTAR Signature System with Ellips Transversal Ultrasound — Comparison of vision after cataract surgery based on two different types of equipment.
  Arms: Abbott WHITESTAR Signature System
Device: Alcon Infiniti wiht the OZIL Torsional Handpiece — Comparision of vision after cataract surgery based on two different types of equipment.
  Arms: Alcon Infiniti

SUMMARY:
The purpose of this study is to look at the outcomes of your vision after your cataract surgery based on two different types of equipment that will be used during your surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 21 scheduled to undergo bilateral phacoemulsification with implantation of multifocal IOLs.
* Both eyes must have similar degrees of cataract and astigmatism (topographic cylinder difference of <2.00D as well as similar globe axial length as measured by the IOL Master of <0.5mm).
* Visual potential of UCVA 20/25/ or better.
* Clear intraocular media other than cataract.

Exclusion Criteria:

* Clinically relevant differences between eyes in ocular disease or pathology.
* Presence of glaucoma, macular disease, or foveal disease to an asymmetrical degree.
* Asymmetrical use of ocular medications.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Kerry Assil, Beverly Hills, California, United States